CLINICAL TRIAL: NCT04424979
Title: Visual Field Expansion Through Innovative Multi-Periscopic Prism Design
Brief Title: Feasibility Tests for Various Prism Configurations for Visual Field Loss
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts Eye and Ear Infirmary (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Principal Investigator, Alexandra Bowers, Associate Professor, Massachusetts Eye and Ear Infirmary
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: MPP_Feasibility1; R01EY023385 (NIH)
Record Dates: First submitted 2020-06-05; First posted 2020-06-11 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Hemianopia, Homonymous; Tunnel Vision; Visual Field Defect, Peripheral; Visual Field Constriction Bilateral; Visual Field Defect Homonymous Bilateral
Keywords: Visual field expansion; Prisms; Hemianopsia; Tunnel vision; Visual field loss
MeSH Terms: conditions — Hemianopsia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- High power prisms (Experimental): Various configurations of high power prisms will be developed for each individual and custom fit into spectacles lenses.
  Interventions: Device: High power prisms

INTERVENTIONS:
Device: High power prisms — High power prisms designed to shift images from blind areas into portions of the wearer's remaining, seeing, field of vision

SUMMARY:
The investigators will develop and test different configurations of high-power prisms to expand the field of vision of patients with visual field loss to assist them with obstacle detection when walking. The study will involve multiple visits (typically four) to Schepens Eye Research Institute for fitting and testing with the prism glasses. The overall objective is to determine best designs and fitting parameters for implementation in prism devices for future clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Visual field loss, either peripheral field loss or hemianopic field loss
* Visual acuity of at least 20/50 in the better eye
* In sufficiently good health to be able to complete sessions lasting 2-4 hours
* Able to independently walk short distances
* Able to give voluntary, informed consent
* Able to speak English

Exclusion Criteria:

* Any physical or mental impairments, including cognitive dysfunction, balance problems or other deficits that could impair the ability to walk or use the prism spectacles
* A history of seizures in the last 6 months
* Hemispatial neglect (subjects with hemianopic field loss only)

Ages: 7 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-11-06 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Field of view expansion | Through study completion, an average of four months
  Horizontal and vertical extent of the expansion (in degrees) of the field of view

SECONDARY OUTCOMES:
Pedestrian detection rate | Through study completion, an average of four months
  Proportion of pedestrians detected (in simulated walking or simulated driving)

CONTACTS AND LOCATIONS:
Overall Officials: Eliezer Peli, MSc, OD, Study Director — Schepens Eye Research Institute of Massachusetts Eye and Ear
Locations (1):
- Schepens Eye Research Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bowers AR, Manda S, Shekar S, Hwang AD, Jung JH, Peli E. Pilot study of a pedestrian collision detection test for a multisite trial of field expansion devices for hemianopia. Optom Vis Sci. 2024 Jun 1;101(6):408-416. doi: 10.1097/OPX.0000000000002152. PMID 38990239